CLINICAL TRIAL: NCT05649410
Title: Effects of Sleeper Stretch and Mobilization With Movement in Patients With Adhesive Capsulitis
Brief Title: Effects of Sleeper Stretch and Mobilizations With Movement in Patients With Adhesive Capsulitis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: REC -01394 Kiran Azam Khan
Record Dates: First submitted 2022-12-06; First posted 2022-12-14 (Actual); Last update posted 2024-12-17 (Actual); Status verified 2024-12

CONDITIONS: Adhesive Capsulitis
Keywords: pain; sleeper stretch; mobilization with movement; range of motion
MeSH Terms: conditions — Bursitis; Pain | interventions — Movement

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- mobilization with movement and conventional therapy (Experimental): Mobilization with movement for Flexion, Abduction, Internal rotation, external rotation
  Interventions: Other: mobilization with movement and conventional therapy
- sleeper stretch along with conventional therapy (Experimental): IT will be performed with the patient in side lying on the affected side to stabilize the scapula against the table and both the shoulder and elbow flexed to 90°.In this position, passive Internal Rotation is applied to the affected shoulder by the therapist or patients opposite hand.
  Interventions: Other: sleeper stretch along with conventional therapy

INTERVENTIONS:
Other: mobilization with movement and conventional therapy — Mobilization with movement for Flexion, Abduction, Internal rotation, external rotation
  Arms: mobilization with movement and conventional therapy
Other: sleeper stretch along with conventional therapy — it will be performed with the patient in side lying on the affected side to stabilize the scapula against the table and both the shoulder and elbow flexed to 90°.In this position, passive Internal Rotation is applied to the affected shoulder by the therapist or patients opposite hand.
  Arms: sleeper stretch along with conventional therapy

SUMMARY:
Adhesive capsulitis is a condition characterized by progressive declination range of motion at the glenohumeral joint due to tightness of capsule. The joint capsule and its surrounding connective tissue becomes stiffed, inflamed and shortened which in return causes decrease in range of motion that progress to chronic pain and stiffness. Adhesive capsulitis is a self-limiting disorder that resolves within 1-3 years.

DETAILED DESCRIPTION:
Idiopathic (primary) adhesive capsulitis occurs spontaneously without a specific precipitating event. Primary adhesive capsulitis results from a chronic inflammatory response with fibro elastic proliferation, which may actually be an abnormal response from the immune system. Secondary adhesive capsulitis occurs after a shoulder injury or surgery or may be associated with another condition such as diabetes, rotator cuff injury, cerebrovascular accident or cardiovascular disease, which may prolong recovery and limit outcomes The prevalence of adhesive capsulitis is estimated at 2% to 5% of the general population. Frozen shoulder mainly affects individuals of 40-65 years of age with a female predominance. Adhesive Capsulitis follows a capsular pattern where external rotation is greatly restricted followed by abduction and internal rotation. Adhesive capsulitis is classically characterized by three stages. The length of each stage is variable, but typically the first stage (freezing) lasts for 3 to 6 months, the second stage (frozen) from 3 to 18 months and the final stage (thawing) from 3 to 6 months Currently various techniques are used, such as the application of moist heat, strengthening exercises, stretching and manual exercises for the treatment of Adhesive Capsulitis .Manual therapy techniques such as high and low grade glenohumeral mobilizations ,Proprioceptive neuromuscular facilitation techniques, Muscle energy Techniques, Mobilization with movement, and Sleeper stretch all have been proved effective for the treatment of adhesive capsulitis through different researches. Conservative treatment includes various exercises method and physical therapy modalities such as a heat therapy, transcutaneous electrical nerve stimulation (TENS), Ultrasound (US), Acupuncture and (Light Amplification by Stimulated Emission of Radiation) LASER

ELIGIBILITY:
Inclusion Criteria:

* Patients with Adhesive Capsulitis of stage 1 and 2.
* Patients with idiopathic adhesive capsulitis.
* Patients with unilateral involvement having painful stiff shoulder for 3 or more months without any shoulder trauma.
* Marked loss in active and passive Range of Motion (Abduction, external and internal rotation) minimum 50% compared to the unaffected side.
* 1.5cm asymmetry on bilateral comparison during lateral scapular slide test.

Exclusion Criteria:

* Patients with shoulder pain due to neurological abnormalities e.g. Hemiplegia.
* Patients with Rotator cuff injury or tear.
* Recent trauma to upper limb.
* Disorders of bones such as fractures, osteoporosis, glenohumeral arthritis.
* Cervical spondylosis or cervical radiculopathy.
* Any malignancy or tumor.
* Patients having any intra articular injection in the gleno-humeral joint during last three months.
* Patients with cardiovascular impairments

Ages: 40 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 44 (Actual)
Dates: Start 2023-01-01 (Actual); Primary Completion 2023-07-10 (Actual); Study Completion 2023-07-10 (Actual)

PRIMARY OUTCOMES:
NPRS (Numeric Pain Rating Scale) | four weeks
  The Numeric Pain Rating Scale (NPRS) measures the subjective intensity of pain. The NPRS is an eleven-point scale from 0 to 10. "0" = no pain and "10" = the most intense pain imaginable. intraclass correlation coefficient = 0.74 for shoulder pain.
Goniometer | four weeks
  Shoulder range of motion i.e. Shoulder Flexion, Extension, Abduction, Adduction, Internal rotation, External rotation will be measured using goniometer, intraclass correlation coefficient for using goniometer for shoulder joint Range Of Motion ranges from 0.91 to 0.99
SPADI (Shoulder Pain and Disability Index) | four weeks
  The Shoulder Pain and Disability Index (SPADI) is a patient completed questionnaire with 13 items assessing pain level and extent of difficulty with Activities of Daily Livings requiring the use of the upper extremities. The pain subscale has 5-items and the Disability subscale has 8-items. The patient is instructed to choose the number that best describes their level of pain and extent of difficulty using the involved shoulder. The pain scale is summed up to a total of 50 while the disability scale sums up to 80. The total SPADI score is expressed as a percentage. A score of 0 indicates best 100 indicates worst. A higher score shows more disability. SPADI is reliable for subjects with Adhesive capsulitis, intraclass correlation coefficient for pain scale=0.989 and intraclass correlation coefficient for disability=0.990
Scapulohumeral Rhythm | four weeks
  Scapular upward rotation will be measured using inclinometer placed at the spine of scapula. Patient will be advised to perform shoulder abduction and measurements will be taken at 3 degrees i.e. 0 to 45degree, 0 to 90 degree, 0 to 120 degree. 3 measurements will be taken at each range and then their mean will be calculated. Scapulohumeral rhythm will be measured by dividing humeral elevation with scapular upward rotation. Scapulohumeral rhythm=humeral elevation/scapular upward rotation. The intraclass correlation coefficient for measuring Scapulohumeral rhythm using inclinometer is > 0.892.

CONTACTS AND LOCATIONS:
Overall Officials: maria Khalid, MSOMPT, Principal Investigator — Riphah International University
Locations (1):
- The Physiotherapy clinic Saidpur Road, Rawalpindi, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No